CLINICAL TRIAL: NCT02506491
Title: A Pilates Exercise Program for Improving Core Strength, Balance and Functional Autonomy in Aged Women: Study Protocol for a Randomized Controlled Trial
Brief Title: A Pilates Exercise Program for Improving Core Strength, Balance and Functional Autonomy in Aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Maria Carrasco, PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMAFI/24/14
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Healthy Aged Women
MeSH Terms: interventions — Exercise Movement Techniques; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pilates exercise program (Experimental): Incorporate Pilates principles to stimulate core muscles in a dynamic and static way, and exercising arms and legs complementarity with balance as an essential part of standing exercises.
  Interventions: Other: Pilates exercise
- Muscular exercise program (Experimental): To train core muscles in a dynamic and static way, and exercising arms and legs complementarity with balance as an essential part of standing exercises.
  Interventions: Other: Muscular exercise
- Control group (Active Comparator): Healthy active but nonexercising old women
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Pilates exercise — 2 sessions/week, 1 hour/session during 18 weeks. Intensity determined from 6 to 9 points, controlled by the Resistance exercise scale of perceived exertion (OMNI-RES).
  Arms: Pilates exercise program
Other: Muscular exercise — 2 sessions/week, 1 hour/session during 18 weeks. Intensity determined from 6 to 9 points, controlled by the Resistance exercise scale of perceived exertion (OMNI-RES).
  Arms: Muscular exercise program
Other: Control Group — No exercise
  Arms: Control group

SUMMARY:
This study is based on assess and contrast isometric and isokinetic core strength, static and dynamic balance, the number of falls, and functional autonomy in three different old women groups after a 18 weeks 1) Pilates-based structured exercise program, 2) muscular structured exercise program, and 3) nonexercising.

DETAILED DESCRIPTION:
Real life conditions require concurrent attention-demanding tasks, increasing the risk of falling and contributing to disability. Pilates-based exercise is proposed as a combined core and mental training program grounded on learning functionally effective postural sets and motor patterns, that will provide better results than a muscular exercise program in old women trunk strength, the risk of falling, functional autonomy and other complementary physical and mental functions. This is a 30-weeks quasi-experimental randomized controlled trial in which 80 independent old women will be allocated to a Pilates-based exercise program, a muscular exercise program, and a no-exercise control group. The intervention is divided into 18 weeks of supervised exercise and a 12 weeks follow-up. Primary outcome will be isokinetic and isometric trunk and hip flexion-extension strength, static and dynamic balance, the number of falls, and functional autonomy. Secondary outcome will include body composition, habitual physical activity and a standardized gerontological evaluation composed of body composition, daily physical activity, the independence to develop basic and instrumental activities of daily living, and the cognitive, affective and social function assessment. Every item will be measured at baseline, 18 and 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 60 to 80 years, physically and mentally able to enroll in the exercise programs. The level of education, toxic habits, medical treatment and/or diseases that can affect musculoskeletal or cardiovascular systems, mental illness, urinary incontinence, the presence of oedema and high blood pressure will be controlled.

Exclusion Criteria:

* Current or prior participation in a structured Pilates-based or muscular exercise program in the past 3 months, and visual or auditory impairments not corrected with glasses or hearing aid. Each participant will also be at least 80% compliant to the exercise.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in trunk and hip isokinetic and isometric muscular flexion/extension peak torque, given in Newtons per meter. | "Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks"
  assessed on a Biodex System III Pro Isokinetic Dynamometer (Biodex Medical System, NY, USA).

SECONDARY OUTCOMES:
Changes in displacement of the center of pressure (millimeters) and time spent standing on two feet, tandem and monopodal display. | Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks"
  assessed with a portable force platform (Kistler, 9286AA).
Changes in time spent to accomplish the Timed Up and Go test for dynamic balance | "Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks"
  participants will be given instructions to stand up from a chair, walk 3 meters as quickly and safely as possible, turn around a cone, walk back and sit down.
number of falls | participants will be followed every 4 weeks
  number of falls registration
Changes in time to accomplish the protocol GDLAM for assessing functional autonomy | Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks
  protocol GDLAM consists of: 10 meters walking speed, standing up from a chair during 5 times, get up the floor from the ventral decubitus position, standing up from a chair and walk around a triangular circuit, and putting on and taking off a T-shirt.
Changes in bone mineral, lean mass (nonbone), and fat mass for total body, head, chest, trunk, hip, right and left legs and arms regions. | "Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks"
  assessed with a dual-energy X-ray bone densitometry (XR-46, Norland Corp., Fort Atkinson, USA).
Changes in score from the Physical Activity Scale for the Elderly (PASE) to measure habitual physical activity. | "Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks"
  The PASE is comprised of self-reported occupational, household and leisure items over a one-week period.
Changes in the Katz scale index to assess the independence to develop basic activities of daily living | "Changes from baseline at 18 weeks" and "Changes from baseline at 30 weeks"
  It summarizes performance in six functions: namely, bathing, dressing, going to toilet, transferring, continence and feeding.
Changes in the Lawton and Brody's scale index to assess the independence to develop instrumental activities of daily living | "Changes from baseline at 22 weeks" and "Changes from baseline at 34 weeks"
  It encomprises eight functional abilities, such as the use of the telephone, shopping, food preparation, housekeeping, laundry, mode of transport, taking medication and handling finances.
Changes in the Mini-Mental State score to assess the cognitive function | "Changes from baseline at 22 weeks" and "Changes from baseline at 34 weeks"
  It covers orientation, memory, attention, calculation, recall and language
Changes in the Geriatric Depression Scale of Yesavage (GDSy) score to determine the affective function | "Changes from baseline at 22 weeks" and "Changes from baseline at 34 weeks"
  It is composed of 15 questions that cover a wide variety of topics relevant to depression, such as somatic complaints, cognitive complaints, motivations, future/past orientation, self-image, losses, agitation, obsessive traits, and mood itself.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carrasco, PhD, Study Director — Universidad de Almeria; Domingo J Ramos-Campo, PhD, Principal Investigator — Universidad Católica San Antonio. Murcia; Jacobo A Rubio-Arias, PhD, Principal Investigator — Universidad Católica San Antonio. Murcia; Delia Reche-Orenes, PhD student, Principal Investigator — Universidad Católica San Antonio. Murcia

REFERENCES:
- [Result] Carrasco M, Martínez I, Vaquero M. Cambios en la fuerza isométrica de las mujeres postmenopáusicas tras el ejercicio en el medio acuático. Revista Internacional de Medicina y Ciencias de la Actividad Física y el deporte 13(49): 73-85, 2013
- [Result] Zaragoza AB, Carrasco M. Condición Física y estado de salud mental en mujeres mayores físicamente independientes. European Journal of Investigation in Health, Psychology and Education. 4(3): 289-300, 2014.
- [Result] Carrasco M, Vaquero M. Training in a shallow pool: Its effect on upper extremity strength and total body weight in postmenopausal women. International SportMed Journal 12(1): 17-29, 2011
- [Result] Carrasco M, Vaquero M. Water training in postmenopausal women: effect on muscular strength. European Journal of Sport Science 12(2): 193-200, 2011
- [Result] Carrasco M, Reche D, Torres-Sobejano M, Romero E, Martínez I. Comparación de la movilidad del raquis entre mujeres de mediana edad practicantes de pilates y de otro tipo de ejercicio. Journal of Sport and Health Research 6(2): 169-176, 2014
- [Result] González-Galvez N, Carrasco M, Marcos-Pardo PJ, Feito Y. The effect of Pilates Method in scholar's trunk strength and hamstring flexibility. Gender differences. International Journal of Medical, Health, Pharmaceutical and Biomedical Engineerin 8(6): 348-351, 2014.
- [Result] Carrasco M, Martínez I, Navarro MD. Daily physical activity and bone mineral density in older women. Revista Brasileira de Medicina do Esporte 21(1): 22-26, 2015.
- [Derived] Carrasco-Poyatos M, Ramos-Campo DJ, Rubio-Arias JA. Pilates versus resistance training on trunk strength and balance adaptations in older women: a randomized controlled trial. PeerJ. 2019 Nov 14;7:e7948. doi: 10.7717/peerj.7948. eCollection 2019. PMID 31741786
- [Derived] Carrasco-Poyatos M, Rubio-Arias JA, Ballesta-Garcia I, Ramos-Campo DJ. Pilates vs. muscular training in older women. Effects in functional factors and the cognitive interaction: A randomized controlled trial. Physiol Behav. 2019 Mar 15;201:157-164. doi: 10.1016/j.physbeh.2018.12.008. Epub 2018 Dec 8. PMID 30529737